CLINICAL TRIAL: NCT02323165
Title: A New Method for Detection of Bacteria in the Bloodstream
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201401005
Record Dates: First submitted 2014-12-11; First posted 2014-12-23 (Estimated); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Burns; Wounds
MeSH Terms: conditions — Burns; Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Burns and Wound Care: Blood samples will be taken to detect and identify a molecular detection of bacteria in the bloodstream. In addition, data will be collected from the standard of care blood samples and compared.
  Interventions: Other: Molecular Detection of Bacteria in the Bloodstream

INTERVENTIONS:
Other: Molecular Detection of Bacteria in the Bloodstream — Extracted nucleic acid will be tested by Polymerase Chain Reaction (PCR) with universal bacterial 16 S amplifiers from known 16 S sequences that routinely contaminate reagents. Polymerase Chain Reaction (PCR) will be performed with both TaqMan assays to provide quantitative copy numbers, as well as traditional PCR that can produce products that can be sequenced to confirm bacterial species identification.

SUMMARY:
The primary aim is to determine if this new technique will detect and identify bacteria in the blood sooner than standard blood cultures or identify patients who may be septic without growing bacteria in their cultures. These will be correlated with the data collected from medical records on presumed sepsis. These results will be linked to data concerning infection that will be available as part of routine care including blood counts and other laboratory values that would be part of the routine medical care such as a white blood cell count. The earlier the bacteria are identified and the appropriate antimicrobials are administered the better the patient outcome.

DETAILED DESCRIPTION:
This study will involve additional blood samples to be taken during the routine clinical blood draw, while the subject is being treated for their burn/wounds. The additional research samples will be examined for bacteria. A second blood draw will be performed at approximately 24 hours of initial blood collection. The blood is being collected and then correlate with results of routine medical care blood cultures and clinical status of the subject (diagnosis of sepsis, hemodynamic instability). Data that will be abstracted from the current electronic medical record includes whether there is any type of catheter indwelling (brand name and type), insertion methods including place of insertion (Intensive Care Unit, Operating Room, Emergency Department), adherence to bundle, complications during insertion, colonization of the subject with bacteria (MRSA), and culture results obtained as part of clinical care. Demographics (subject's age) and diagnoses will also be captured as some studies have shown a higher risk of infection with certain processes (burns) and percentage of burn.

ELIGIBILITY:
Inclusion Criteria:

* Burn patient with ≥20 % total body surface area burns or non-burned wound care patient requiring wound care in the Burn Intensive Care Unit.
* Must weigh ≥ 50 kilograms

Exclusion Criteria:

* Pregnant or Lactating women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Identification of potential patients will take place during normal medical care of burn and wound patients admitted to the Burn Intensive Care Unit.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of new molecular technique for the detection of bacteria in the blood stream. (Extracted nucleic acid will be tested by PCR) | 6 months
  Extracted nucleic acid will be tested by PCR with "universal" bacterial 16 S primers that we have identified as not amplifying a product from known 16 S sequences that routinely contaminate reagents.PCR will be performed by both TaqMan assays we have developed that can provide quantitative copy numbers, as well as traditional PCR that can produce products that can be sequenced to confirm bacterial species identification.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Fahy, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Department of Anesthesia and Critical Care, Department of Surgery, Department of Pathology, Immunology and Laboratory Medicine in conjunction with UF Health at Shands Hosptial at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No